CLINICAL TRIAL: NCT04122963
Title: CLOSE-guided Pulmonary Vein Isolation Using High Power and Stable RF Applications: a Randomized Study. The POWERAF Study
Brief Title: CLOSE-guided Pulmonary Vein Isolation Using High Power and Stable RF Applications
Acronym: POWERAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Sebastien Knecht, Professor Doctor, AZ Sint-Jan AV
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2406
Record Dates: First submitted 2019-10-09; First posted 2019-10-10 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High power group (Active Comparator): The experimental group will receive AF ablation with 45 Watt and stricter stability criteria (3 mm for 3 seconds).
  Interventions: Procedure: High power CLOSE-guided PVI ablation
- Standard group (Active Comparator): The control group will receive AF ablation according to the standard CLOSE-protocol (35 Watt and stability criteria of 3 mm for 8 seconds)
  Interventions: Procedure: Standard CLOSE-guided PVI ablation

INTERVENTIONS:
Procedure: High power CLOSE-guided PVI ablation — CLOSE-guided PVI ablation with 45 Watt and stricter stability criteria (3 mm for 3 seconds)
  Arms: High power group
Procedure: Standard CLOSE-guided PVI ablation — Standard AF ablation according to the CLOSE-protocol
  Arms: Standard group

SUMMARY:
In this prospective, randomised, controlled, unblinded,monocentric study, we aim to evaluate the safety and efficacy of higher power CLOSE-guided PVI in patients referred for a first ablation for paroxysmal AF. We aim to include 100 patients into two groups (1:1). The experimental group will receive AF ablation with 45 Watt and stricter stability criteria (3 mm for 3 seconds) compared to the control group which will receive AF ablation according to the standard CLOSE-protocol (35 Watt and stability criteria of 3 mm for 8 seconds).

DETAILED DESCRIPTION:
BACKGROUND: In a population of paroxysmal AF 'CLOSE'-guided PVI (Target Ablation index (AI) >550 and >400 for anterior and posterior wall respectively, interlesion distance ≤6mm) has been shown to obtain single-procedure durable PV isolation. However, the optimal RF power and stability criteria is unknown.

OBJECTIVES: With this study, we aim at evaluation the efficacy and the safety of higher power (45 watts) and stricter stability criteria (3 mm for 3 sec) as compared to a standard CLOSE protocol (35 watts with stability of 3 mm for 8 sec) in patients referred for a first ablation for paroxysmal AF.

POPULATION: Eligible patients are patients with paroxysmal AF who are planned for a 'CLOSE'-guided PV isolation for paroxysmal AF. At the time of the procedrual planning, we will ask the patient his/her consent for collectio of data. We aim at including 100 patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred for symptomatic paroxysmal AF and without advanced structural heart disease
* Signed Patient Informed Consent Form
* Age 18 years or older
* Able and willing to comply with all follow-up testing and requirements

Exclusion Criteria:

* Persistent atrial fibrillation (history of AF>7days or history of cardioversion > 48h of AF)
* Previous ablation for AF
* LA antero-posterior diameter>50 mm (parasternal long axis view , PLAX)
* LVEF <35% (ejection fraction)
* AF secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause
* CABG procedure within the last three months
* Awaiting cardiac transplantation or other cardiac surgery
* Documented left atrial thrombus on imaging
* Diagnosed atrial myxoma
* Women who are pregnant or breastfeeding
* Acute illness or active systemic infection or sepsis
* Unstable angina
* Uncontrolled heart failure
* Myocardial infarction within the previous two months
* History of blood clotting or bleeding abnormalities
* Contraindication to anticoagulation therapy (ie, heparin or warfarin)
* Life expectancy less than 12 months
* Enrollment in any other study evaluating another device or drug
* Presence of intramural thrombus, tumor or other abnormality that precludes catheter introduction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Efficacy: Acute procedural success | At time of ablation
  First pass pulmonary vein isolation confirmed after adenosine injection
Safety: Absence of clinical complications | From time of ablation to 1 month post procedure
  Absence of clinical complications during the procedure and up to one month thereafter

SECONDARY OUTCOMES:
Procedural duration time | At time of ablation
Duration for pulmonary vein isolation | At time of ablation
Fluoroscopic duration and irradiation (AK) | At time of ablation
Amount of ablation points associated with temperature rise | At time of ablation
Maximum temperature in case of temperature rise | At time of ablation
Incidence of adverse events related to ablation | From time of ablation to 6 months post procedure
First pass encirclement isolation rate | At time of ablation
Reconnection rate after adenosine | At time of ablation
Number of dislocations | At time of ablation
Number of ablation points with an oesophageal temperature rise >39°C | At time of ablation
Maximum temperature in case of oesophageal temperature rise | At time of ablation
Longterm procedural success rate | Six months after ablation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Bruges, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wielandts JY, Kyriakopoulou M, Almorad A, Hilfiker G, Strisciuglio T, Phlips T, El Haddad M, Lycke M, Unger P, Le Polain de Waroux JB, Vandekerckhove Y, Tavernier R, Duytschaever M, Knecht S. Prospective Randomized Evaluation of High Power During CLOSE-Guided Pulmonary Vein Isolation: The POWER-AF Study. Circ Arrhythm Electrophysiol. 2021 Jan;14(1):e009112. doi: 10.1161/CIRCEP.120.009112. Epub 2020 Dec 10. PMID 33300809